CLINICAL TRIAL: NCT00223106
Title: A Prospective Multicenter Clinical Study on a New Approach in Treating Stress and Mixed Incontinence and Vaginal Vault Prolapse
Brief Title: Treatment for Stress and Mixed Urinary Incontinence and Vaginal Vault Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: WHC03001
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Urinary Incontinence, Stress; Mixed Incontinence; Vaginal Vault Prolapse
Keywords: urge incontinence; urinary incontinence; vault prolapse; stess incontinence; mixed incontinence; urine leakage; enterocele; rectocele; cystocele
MeSH Terms: conditions — Urinary Incontinence, Stress; Pelvic Organ Prolapse; Urinary Incontinence, Urge; Urinary Incontinence; Hernia; Rectocele; Cystocele | interventions — Suburethral Slings

INTERVENTIONS:
Device: Vaginal Sling

SUMMARY:
The primary objective of this study is to further evaluate the safety and effectiveness of the use of a sling device in women for stress and mixed urinary incontinence as well as vaginal vault prolapse.

DETAILED DESCRIPTION:
Urinary incontinence is the involuntary loss of urine and can affect both men and women throughout their lives. Women are more likely to develop incontinence as a result of pregnancy and childbirth. There are approximately 11 million cases of incontinence in the US contributing to several different types of incontinence including :

* Urge - 30% of the market
* Stress - 30% of the market of which 85% are women
* Combination urge and stress - 40%

Despite advances in behavioral therapy, pharmacological advances as well as development of minimally invasive surgical procedures, only one out of every twelve people affected actually seek help.

Prolapse

Globally, approximately 1 million women suffer uterovaginal prolapse annually and this condition can be associated with urinary incontinence. The breakdown of treatments for uterovaginal prolapse includes:

* 20% - no treatment
* 20% - non surgical management (pessary)
* 60% - receive a surgical procedure of a suture repair or mesh repair

There were greater than 600,000 surgeries performed globally to treat prolapse. These numbers are projected to increase due to rapid, easy, and less costly methods as well as new products that facilitate the easier procedures.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be female and >18 years of age.
* Subject must have genuine stress or mixed incontinence AND/OR evidence of pelvic organ prolapse.

Exclusion Criteria:

* Any subject with clotting defects, bleeding disorders or receiving anticoagulant treatments AND is determined to be at risk for minimally invasive surgery as determined by the investigator
* Subjects who currently have an untreated urinary tract infection
* Subject is unable to comply with the study requirements, follow-up schedule, or to give valid informed consent.
* Subject is pregnant or desires future pregnancies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2004-03; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy for incontinence and prolapse procedures.

SECONDARY OUTCOMES:
Quality of Life Improvement as determined by Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Noreen A. Gannon, Study Director — Medtronic - MITG
Locations (1):
- US Surgical, Norwalk, Connecticut, United States